CLINICAL TRIAL: NCT06424184
Title: Substance Use Disorder Treatment With Accelerated Repetitive Transcranial Magnetic Stimulation for Depression (START-D)
Brief Title: Accelerated rTMS for Substance Use Disorder and Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Manish Jha, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2024-0232
Record Dates: First submitted 2024-05-10; First posted 2024-05-22 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Stimulant Use; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Open label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- rTMS Intervention (Experimental): Eligible participants who are enrolled will receive an accelerated course of repetitive Transcranial Magnetic Stimulation.
  Interventions: Device: Accelerated Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Accelerated Repetitive Transcranial Magnetic Stimulation — The rTMS protocol implemented in this study will include approximately 10-minute long sessions of intermittent theta burst stimulation (iTBS) with at least 50 minutes in between iTBS sessions.
  Study participants will receive the rTMS intervention for up to 50 sessions across a three-week period. The total of 50 sessions will be administered as up to 4 sessions each day, up to 5 days per week over an up to 3-week-long period.

SUMMARY:
This study is a small open-label feasibility trial of an accelerated course of repetitive transcranial magnetic stimulation (rTMS) for individuals with depression and stimulant use disorder [including methamphetamine or cocaine use disorder (MUD/CUD)].

DETAILED DESCRIPTION:
This research is an open label feasibility trial of accelerated course of repetitive transcranial magnetic stimulation (rTMS) for individuals with stimulant use disorder. Participants will be recruited from an existing and ongoing longitudinal study of stimulant use disorder (STIM-RAD) (NCT06073340). Prior to initiating the accelerated course of rTMS, participants will undergo screening procedures to evaluate eligibility. Those eligible will complete up to four (4) rTMS sessions of intermittent theta burst over left dorsolateral prefrontal cortex per day, up to five (5) days per week of the study, for a total of 50 sessions over a three (3) week period and will undergo electroencephalography (EEG), electrocardiography (ECG), urine drug screens, as well as self-report and clinician-rated assessments. A follow-up visit will be conducted 1 week after the last session of rTMS.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged 18-65 years, inclusive.
2. Be able to sufficiently understand, speak, and read English to provide informed consent and ask relevant questions, and be willing to comply with all study procedure instructions.
3. Self-report stimulant use (cocaine, methamphetamine, or prescription stimulants) at least 10 days in the 30-day period prior to consent.
4. Have a diagnosis of moderate or severe Cocaine or Methamphetamine Use Disorder (CUD/MUD) or other Stimulant Use Disorder over the past 12 months (as determined by the MINI International Neuropsychiatric Interview).
5. Have a PHQ9 of greater than or equal to five (5).
6. Be willing to provide urine samples, EEGs, and ECGs.
7. Be willing to use appropriate birth control method during the treatment phase of the study, if individual is of childbearing potential.

Exclusion Criteria:

1. Have a current pattern of alcohol, benzodiazepine, or other sedative/hypnotic use that would preclude safe participation in the study, as determined by the PI or their designee.
2. Have a history of a serious medical disorder that, in the opinion of the PI or their designee, would make it unsafe to participate in the study or may prevent collection of study data (e.g., disabling terminal diagnosis for which hospice care is being sought; serious illness requiring systemic treatment and/or hospitalization until participant either completes therapy and/or is clinically stable on therapy, in the opinion of the PI or their designee, prior to study entry).
3. Have a documented history of unprovoked seizure (lifetime) or any seizure in the past 6 months.
4. Have a documented history of brain lesion(s) and/or tumor(s).
5. Have metal implants or non-removable metal objects above the neck.
6. Current pregnancy as determined by a urine screening.
7. Current or lifetime manic or hypomanic episode, defined by MINI diagnostic interview.
8. Current psychotic disorder.
9. Are a prisoner or in police custody at the time of eligibility screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of an accelerated course of repetitive Transcranial Magnetic Stimulation (rTMS). | 3 weeks
  Feasibility will be measured by completion of at least 30 out of 50 sessions of rTMS.

SECONDARY OUTCOMES:
Attainment of response of rTMS intervention on stimulant use assessed by Urine Drug Screens. | 3 weeks
  Attainment of response is defined as 3 out of 5 negative urine samples for stimulants (cocaine, amphetamines), in week 3 of treatment.
Changes in stimulant craving during the 3-week treatment phase assessed by the Stimulant Craving Questionnaire (STCQ). | 3 weeks
  The Stimulant Craving Questionnaire (STCQ) is a 10-item self-report measure derived from the 10-item Cocaine Craving Questionnaire-Brief and the original 46-item Cocaine Craving Questionnaire-Now. The STCQ assesses current craving for stimulants (cocaine, methamphetamine, and other stimulants) using a seven-point scale, with answers ranging from "strongly disagree" to "agree."
Changes in stimulant craving during the 3-week treatment phase assessed by a Visual Analog Drug Craving Scale (VAS). | 3 weeks
  Craving for stimulants and other substances will be self-reported by participants on a Visual Analog Drug Craving Scale (VAS) which ranges from 0 (no craving) to 100 (most intense craving possible).
Changes in stimulant craving during the 3-week treatment phase assessed by the Cue Craving Assessment. | 3 weeks
  Current craving for stimulants will be assessed using the Cue Craving Assessment. Participants will be asked about their current craving for and ability to resist stimulants on a 0-10 scale immediately after cue exposure prior to rTMS and after the completion of each rTMS session. A "0" rating indicates the absence of craving or the absence of the ability to resist use, whereas a "10" rating indicates the highest craving or strongest ability to resist use.
Changes in frequency of self-reported stimulant use based on Timeline Followback (TLFB). | 6 weeks
  The Timeline Followback (TLFB) procedure will be used to elicit the participant's self-reported use of illicit substances, including but not limited to stimulants, and polysubstance use starting at the Screening Visit and continuing throughout study participation. During the Screening Visit, this form will be used to assess illicit use of substances for the 30-day period prior to written consent. During the study, TLFB will be administered to document the participant's self-reported use of illicit substances, nicotine, and tobacco for each visit since the previous TLFB assessment. Participant's drug of choice will be asked and determined by study coordinator and recorded along with the TLFB assessment.
Changes in self-reported symptoms of suicidality during the 3-week treatment phase. | 3 weeks
  The Concise Health Risk Tracking - Self-Report (CHRT-SR) is a 14-item self-report assessment of suicidality and related thoughts and behaviors. The scale is designed to track suicidality quickly and easily in a manner consistent with the Columbia Classification Algorithm of Suicide Assessment (C-CASA). Participants are asked to rate the extent that they have related to fourteen different statements on a scale of "strongly disagree" to "strongly agree." A higher score indicates higher suicidality.
Changes in self-reported symptoms of depression during the 3-week treatment phase. | 3 weeks
  The Quick Inventory of Depressive Symptomatology Self-Report (QIDS-SR) will assess overall depressive symptoms. The total score of QIDS-SR (range of 0-27) is based on the nine Diagnostic and Statistical Manual of Mental Disorders (DSM-lV) criteria symptom domains: sad mood, concentration, self-outlook, suicidal ideation, involvement, energy/fatigability, sleep disturbance, appetite/weight increase/decrease, and psychomotor agitation/retardation. Each question is scored on a 0-3 scale based on the participant's response. A higher score indicates higher depressive symptoms.
Changes in self-reported symptoms of irritability during the 3-week treatment phase. | 3 weeks
  A 10-item version of the Concise Associated Symptom Tracking Scale Self-Report (CAST-IRR) will be used to assess associated mood symptoms. Participants are asked to rate the extent that they have related to ten different statements in the past week on a 5-point Likert scale (from 1, "strongly disagree," to 5, "strongly agree," where a higher score indicates increased symptoms). Some items in the CAST-IRR include: "I wish people would just leave me alone"; "I feel very uptight"; "I find myself saying or doing things without thinking"; "Lately everything seems to be annoying me"; and "I find people get on my nerves easily."

CONTACTS AND LOCATIONS:
Overall Officials: Manish Jha, M.B.B.S, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Northrup TF, Green C, Walker R, Greer TL, Trivedi MH. On the invariance of the Stimulant Craving Questionnaire (STCQ) across cocaine and methamphetamine users. Addict Behav. 2015 Mar;42:144-7. doi: 10.1016/j.addbeh.2014.11.020. Epub 2014 Nov 25. PMID 25462663
- [Background] Wewers ME, Lowe NK. A critical review of visual analogue scales in the measurement of clinical phenomena. Res Nurs Health. 1990 Aug;13(4):227-36. doi: 10.1002/nur.4770130405. PMID 2197679
- [Background] Sobell LC, Sobell MB, Leo GI, Cancilla A. Reliability of a timeline method: assessing normal drinkers' reports of recent drinking and a comparative evaluation across several populations. Br J Addict. 1988 Apr;83(4):393-402. doi: 10.1111/j.1360-0443.1988.tb00485.x. No abstract available. PMID 3395719
- [Background] Trivedi MH, Wisniewski SR, Morris DW, Fava M, Gollan JK, Warden D, Nierenberg AA, Gaynes BN, Husain MM, Luther JF, Zisook S, Rush AJ. Concise Health Risk Tracking scale: a brief self-report and clinician rating of suicidal risk. J Clin Psychiatry. 2011 Jun;72(6):757-64. doi: 10.4088/JCP.11m06837. PMID 21733476
- [Background] Posner K, Oquendo MA, Gould M, Stanley B, Davies M. Columbia Classification Algorithm of Suicide Assessment (C-CASA): classification of suicidal events in the FDA's pediatric suicidal risk analysis of antidepressants. Am J Psychiatry. 2007 Jul;164(7):1035-43. doi: 10.1176/ajp.2007.164.7.1035. PMID 17606655
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Background] Rush AJ, Bernstein IH, Trivedi MH, Carmody TJ, Wisniewski S, Mundt JC, Shores-Wilson K, Biggs MM, Woo A, Nierenberg AA, Fava M. An evaluation of the quick inventory of depressive symptomatology and the hamilton rating scale for depression: a sequenced treatment alternatives to relieve depression trial report. Biol Psychiatry. 2006 Mar 15;59(6):493-501. doi: 10.1016/j.biopsych.2005.08.022. Epub 2005 Sep 30. PMID 16199008
- [Background] Trivedi MH, Wisniewski SR, Morris DW, Fava M, Kurian BT, Gollan JK, Nierenberg AA, Warden D, Gaynes BN, Luther JF, Rush AJ. Concise Associated Symptoms Tracking scale: a brief self-report and clinician rating of symptoms associated with suicidality. J Clin Psychiatry. 2011 Jun;72(6):765-74. doi: 10.4088/JCP.11m06840. PMID 21733477
- [Background] Jha MK, Minhajuddin A, South C, Rush AJ, Trivedi MH. Irritability and Its Clinical Utility in Major Depressive Disorder: Prediction of Individual-Level Acute-Phase Outcomes Using Early Changes in Irritability and Depression Severity. Am J Psychiatry. 2019 May 1;176(5):358-366. doi: 10.1176/appi.ajp.2018.18030355. Epub 2019 Mar 29. PMID 30922100